CLINICAL TRIAL: NCT04173936
Title: Effects of a Community-based Tai Chi Program on Balance, Functional Outcomes, and Sensorimotor Function in Older Adults
Brief Title: Community-based Tai Chi, Balance, and Fall Risk
Status: Completed | Type: Observational
Sponsor: University of North Carolina at Asheville (Other)
Responsible Party: Sponsor
Other Study IDs: 1373542-1
Record Dates: First submitted 2019-11-18; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Postural Balance; Fall; Proprioceptive Disorders
MeSH Terms: conditions — Somatosensory Disorders | interventions — Tai Ji

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tai Chi: All participants enrolled in a 12 week community-based tai chi program.
  Interventions: Behavioral: tai chi

INTERVENTIONS:
Behavioral: tai chi — 12-week community-based tai chi program

SUMMARY:
Aims: Examine the effects of a community Tai Chi program on measures of balance and sensorimotor function.

Methods: In a pre-test and post-test design, balance was measured in older adults (N=344; 73.4±7.4 years) with 30-second chair stand, timed-up and go, and 4-stage balance test following a 12-week community-based tai chi intervention. Balance measures and additional sensorimotor measures, including hip abductor electromechanical delay and hip proprioception, were measured in a smaller sample of older adults (n=11; 67.3±3.7 years).

ELIGIBILITY:
Inclusion Criteria:

* age 60 years or older
* ability to independently ambulate
* self-described concern with stability and/or mobility.

Exclusion Criteria:

* Neurological diagnosis
* Participants body weight exceeds >450 pounds).

Ages: 60 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Older adult volunteers willing to participate in a 12-week community-based tai chi program
Sampling Method: Non-Probability Sample
Enrollment: 405 (Actual)
Dates: Start 2014-01-11 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
30-second chair number | 12 weeks
  The number of times a person can stand up and sit down from a chair in 30 seconds
Timed Up and Go | 12 weeks
  The time (in seconds) for a person to stand from a chair, walk 10 feet, turn 180 degrees and return to sit in the chair
4 stage balance test | 12 weeks
  How long (in seconds) can a person stand with feet together, stand with one foot forward and to the side, stand in tandem (one foot immediately in front of the other, and stand on one foot
Hip abductor muscle contraction time | 12 weeks
  Hip abductor muscle contraction speed as measured as the time (in milliseconds) between the onset of electromyography signal and torque onset from hip muscle abduction
Brief-Balance Evaluation System Test | 12 weeks
  The bBESTest is an 8-item, clinically-based assessment measuring anticipatory postural adjustments, compensatory postural responses, sensory orientation, stability in gait, and the timed up-and-go test.
Activities-Specific Balance Confidence Scale (ABC) scale | 12 weeks
  the ABC scale assesses self-reported confidence during 16 activities related to mobility.
Hip joint proprioception error | 12 weeks
  The magnitude of proprioception error was measured on the participant's dominant lower extremity with a custom-built device25,51 that allows for rotation around the axis of a semi-goniometer to measure proprioception in the transverse plane at the hip joint. Proprioception was assessed by measuring the accuracy of actively pointing a marked line on the second toe to target angles along the semi-goniometer during two conditions, a vision condition and an occluded vision condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Wingert, Phd, Principal Investigator — UNC Asheville
Locations (1):
- UNC Asheville, Asheville, North Carolina, United States